CLINICAL TRIAL: NCT05892991
Title: Influence of Using Different Amplitude Modulated Frequencies on the Effectiveness of Interferential Current in Treating Trapezius Trigger Points: a Randomized Controlled Trial.
Brief Title: Using Different Amplitude-modulated Frequencies of IFC for the Treatment of Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, principal investigator, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2023-289
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-05

CONDITIONS: Trigger Point Pain
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: 4 arms will receive treatment for 4 weeks
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be allocated to groups by a researcher not involved in assessment or treatment (AAI). Permuted blocks generated using http://www.randomization.com/ were used for the allocation to assure equal and random allocation. Randomization codes were kept confidential in sealed opaque envelopes and sequentially numbered to ensure concealed allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- standard physical therapy group (Active Comparator): this group will receive 4 physical therapy sessions per week for 4 weeks. The session will consist of intermittent neuromuscular inhibition which is composed of 3 manual approaches (positional release, muscle energy technique, and progressive pressure release).
  Interventions: Other: interferential current
- amplitude modulated frequency (AMF) 130Hz group (Experimental): 1. Chattanooga (Intellect© Advanced, USA) multi-current device will be used to apply the IFC sessions. Carrier frequency 4000Hz, 2 pole placement (pre-modulated), the intensity will be raised till the patient feels a strong but comfortable tingling sensation, AMFs 130. Two vacuum electrodes of medium size will be placed at both sides of the trigger point. The duration of the session will be 30 minutes and will be repeated 3 times per week for 4 weeks.
  2. standard physical therapy treatment as in the first group
  Interventions: Other: interferential current
- amplitude modulated frequency (AMF) 80Hz group (Experimental): 1. Chattanooga (Intellect© Advanced, USA) multi-current device will be used to apply the IFC sessions. Carrier frequency 4000Hz, 2 pole placement (pre-modulated), the intensity will be raised till the patient feels a strong but comfortable tingling sensation, AMFs 80Hz. Two vacuum electrodes of medium size will be placed at both sides of the trigger point. The duration of the session will be 30 minutes and will be repeated 3 times per week for 4 weeks.
  2. standard physical therapy treatment as in the first group
  Interventions: Other: interferential current
- amplitude modulated frequency 4Hz group (Experimental): 1. Chattanooga (Intellect© Advanced, USA) multi-current device will be used to apply the IFC sessions. Carrier frequency 4000Hz, 2 pole placement (premodulated), the intensity will be raised till muscle twitching is visible under electrodes, AMFs 4 Hz. Two vacuum electrodes of medium size will be placed at both sides of the trigger point. The duration of the session will be 30 minutes and will be repeated 3 times per week for 4 weeks.
  2. standard physical therapy treatment as in the first group
  Interventions: Other: interferential current

INTERVENTIONS:
Other: interferential current — this intervention is a type of therapeutic electrical currents of medium frequency used commonly in physical therapy to relieve acute and chronic pain as well as stimulate muscle contraction.
  Other Names: medium frequency current

SUMMARY:
the authors of this work will conduct a randomized controlled trial intended to examine different amplitude-modulated frequencies of interferential current on different measures related to chronic trigger points located in the upper trapezius muscle.

DETAILED DESCRIPTION:
this randomized controlled trial was designed to fill a gap in the literature regarding the most effective amplitude-modulated frequency of interferential current on pain pressure threshold, cervical ROM, and function of the neck region.

this study will be consisted of 4 groups, all groups will receive standard manual treatment commonly used for the treatment of chronic trigger points. this treatment will be conducted 3 times per week for 4 weeks. The standard treatment will consist of an intermittent neuromuscular inhibition technique.

the 3 experimental groups will receive interferential current sessions (3/week) for 4 weeks with the same parameters except for the amplitude-modulated frequency.

outcome measurements will be assessed at baseline, at 4 weeks, and at 4 weeks of the end of the treatment (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* males or females,
* 17 - 50 years of age,
* unilateral pain in the cervical, neck, and upper shoulder, pain persists for 3 months or more,
* pain should be not less than 2 on the visual analog scale (VAS),
* having positive signs of chronic (latent) trigger point(s) in the upper trapezius muscle

Exclusion Criteria:

* cervical and or shoulder pathologies such as disc lesions, arthritis, or compression problems.
* neurological symptoms in the upper limb such as radiculopathy.
* previous cervical, thoracic, or shoulder surgery.
* regular sports practice.
* heavy work-related activities.
* trauma to the cervical spine (whiplash injury).
* osteoporosis.
* complex regional pain syndrome.
* thoracic outlet syndrome
* regular analgesic drugs.

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Active Range of motion (AROM) for cervical spine. | at baseline
  Active range of motion (AROM) of neck side flexion (ipsilateral and contralateral) will be measured using a valid and reliable inclinometer application for Android phone. Measurements will be collected while the participant seated on a chair with back support. The phone will be placed horizontally on the back of the head while the participants assume neutral head position. The participant will be instructed to keep the shoulder rested and move the head to one side till the end of the available range. The procedure will be repeated 3 times and the average value will be used for analysis.
Active Range of motion (AROM) for cervical spine. | at 4 weeks
  Active range of motion (AROM) of neck side flexion (ipsilateral and contralateral) will be measured using a valid and reliable inclinometer application for Android phone. Measurements will be collected while the participant seated on a chair with back support. The phone will be placed horizontally on the back of the head while the participants assume neutral head position. The participant will be instructed to keep the shoulder rested and move the head to one side till the end of the available range. The procedure will be repeated 3 times and the average value will be used for analysis.
Active Range of motion (AROM) for cervical spine. | at 4 weeks after the end of the treatment (follow-up)
  Active range of motion (AROM) of neck side flexion (ipsilateral and contralateral) will be measured using a valid and reliable inclinometer application for Android phone. Measurements will be collected while the participant seated on a chair with back support. The phone will be placed horizontally on the back of the head while the participants assume neutral head position. The participant will be instructed to keep the shoulder rested and move the head to one side till the end of the available range. The procedure will be repeated 3 times and the average value will be used for analysis.
Pain pressure threshold by pressure algometer | at baseline
  The assessor will assess the pain pressure threshold in Kg/cm2 using a pressure algometer (FDIX25 Digital Force Gauge, Greenwich, CT, USA). The algometer will be placed with its tip perpendicular over the TrP then gradual pressure will be applied. The participants will be asked to report pain once they feel it. Measurements will be repeated twice with 30-s rest intervals in-between trials. The mean value will be used for analysis. the more improvement the higher value of pain pressure can be tolerated before pain sensation percieved
Pain pressure threshold by pressure algometer | at 4 weeks
  The assessor will assess the pain pressure threshold in Kg/cm2 using a pressure algometer (FDIX25 Digital Force Gauge, Greenwich, CT, USA). The algometer will be placed with its tip perpendicular over the TrP then gradual pressure will be applied. The participants will be asked to report pain once they feel it. Measurements will be repeated twice with 30-s rest intervals in-between trials. The mean value will be used for analysis. the more improvement the higher value of pain pressure can be tolerated before pain sensation percieved
Pain pressure threshold by pressure algometer | at 4 weeks after the end of the treatment (follow-up)
  The assessor will assess the pain pressure threshold in Kg/cm2 using a pressure algometer (FDIX25 Digital Force Gauge, Greenwich, CT, USA). The algometer will be placed with its tip perpendicular over the TrP then gradual pressure will be applied. The participants will be asked to report pain once they feel it. Measurements will be repeated twice with 30-s rest intervals in-between trials. The mean value will be used for analysis. the more improvement the higher value of pain pressure can be tolerated before pain sensation percieved
Function using neck disability index | at baseline
  The participant's functional status will be assessed by a validated Arabic version of the neck disability index (NDI). The NDI is a 10-item questionnaire scored from 0-50 points (0-100%) in which higher scores indicate higher levels of disability. The cutoff points are: score of 5-14 points (10- 28%) indicates mild disability, 15-24 points (30-48%) indicates moderate disability, 25-38 points (50-68%) indicates severe disability, and above 34 points (68%) for complete disability
Function using neck disability index | at 4 weeks
  The participant's functional status will be assessed by a validated Arabic version of the neck disability index (NDI). The NDI is a 10-item questionnaire scored from 0-50 points (0-100%) in which higher scores indicate higher levels of disability. The cutoff points are: score of 5-14 points (10- 28%) indicates mild disability, 15-24 points (30-48%) indicates moderate disability, 25-38 points (50-68%) indicates severe disability, and above 34 points (68%) for complete disability
Function using neck disability index | at 4 weeks after the end of treatment (follow-up)
  The participant's functional status will be assessed by a validated Arabic version of the neck disability index (NDI). The NDI is a 10-item questionnaire scored from 0-50 points (0-100%) in which higher scores indicate higher levels of disability. The cutoff points are: score of 5-14 points (10- 28%) indicates mild disability, 15-24 points (30-48%) indicates moderate disability, 25-38 points (50-68%) indicates severe disability, and above 34 points (68%) for complete disability
number of painful episode in the trapezius muscle | at baseline
  This outcome will be simply assessed by asking the participant try to accurately determine the number of pain attacks in the affected muscle during the last/ previous 4 weeks. the participant will report the number of painful episodes during the last 4 weeks before engaging in the study, then at the 4 months of the treatment program, then at 4 weeks of the end of the treatment program
number of painful episode in the trapezius muscle | at 4 weeks
  This outcome will be simply assessed by asking the participant try to accurately determine the number of pain attacks in the affected muscle during the last/ previous 4 weeks. the participant will report the number of painful episodes during the last 4 weeks before engaging in the study, then at the 4 months of the treatment program, then at 4 weeks of the end of the treatment program
number of painful episode in the trapezius muscle | at 4 weeks after the end of treatment (follow-up)
  This outcome will be simply assessed by asking the participant try to accurately determine the number of pain attacks in the affected muscle during the last/ previous 4 weeks. the participant will report the number of painful episodes during the last 4 weeks before engaging in the study, then at the 4 months of the treatment program, then at 4 weeks of the end of the treatment program

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Hisham Hussein, Hail, Ha'il Region
  - University of Hail, Hail, Ha'il Region

IPD SHARING:
Plan to Share IPD: No
all data will be with the principal investigator